CLINICAL TRIAL: NCT03018366
Title: Atherosclerosis, Immune Mediated Inflammation and Hypoestrogenemia in Young Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Chrisandra Shufelt, Professor and Chair, Division of General Internal Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO26081
Record Dates: First submitted 2016-12-01; First posted 2017-01-12 (Estimated); Results first posted 2025-02-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Estrogen Deficiency; Cardiovascular Disease (CVD); Functional Hypothalamic Amenorrhea; Endothelial Dysfunction
Keywords: estrogen; premenopause; menopause; amenorrhea
MeSH Terms: conditions — Cardiovascular Diseases; Amenorrhea | interventions — Estradiol; Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 17Beta Estradiol, Progesterone (Active Comparator): 17Beta Estradiol (0.1mg/day) , Progesterone (100mg) or Medroxyprogesterone (10mg) for patient with a peanut allergy because progesterone 100mg is a peanut based product
  Interventions: Drug: 17beta Estradiol; Drug: Progesterone
- Transdermal Placebo Patch, Placebo Pill (Placebo Comparator): Placebo Transdermal Patch, Placebo Pill
  Interventions: Drug: Transdermal placebo patch; Drug: Placebo Pill

INTERVENTIONS:
Drug: 17beta Estradiol — Participants will use a dose of transdermal estradiol 0.1 mg/day patch for 12 weeks +/- 1week. PAT index vascular measures and serum immune markers will be measured after 6 and 12 weeks +/- 1week on estrogen patches. Patches will be applied by the participant to the lower abdomen twice weekly, alternating sides.
  Other Names: Estradiol Transdermal Patch; Vivelle-Dot
  Arms: 17Beta Estradiol, Progesterone
Drug: Transdermal placebo patch — Participants will use a dose of placebo patches for 12 weeks +/- 1 week. Placebos will be applied by the participant to the lower abdomen twice weekly, alternating sides.
  Arms: Transdermal Placebo Patch, Placebo Pill
Drug: Progesterone — After 12 weeks +/- 1week of transdermal estradiol patch, participants will use estrogen patch plus progesterone for 2 additional weeks +/- 3 days. Progesterone is a peanut based product and for patients with a peanut allergy we will replace this with a synthetic progestin at an equivalent dose, medroxyprogesterone 10mg.
  Other Names: Prometrium
  Arms: 17Beta Estradiol, Progesterone
Drug: Placebo Pill — After 12 weeks +/- 1week of transdermal placebo patch, participants will use placebo patch plus placebo pill for 2 additional weeks +/- 3 days.
  Other Names: Placebo Oral Pill
  Arms: Transdermal Placebo Patch, Placebo Pill

SUMMARY:
The purpose of this study is to determine whether young women with functional hypothalamic amenorrhea (premenopausal HypoE) is associated with risk factors for pre-clinical cardiovascular disease (CVD).

For this study, the investigators will measuring vascular function and inflammatory markers on:

* young women with functional hypothalamic amenorrhea (>3 months of no menstrual cycle due to low estrogen)
* young women with regular menstrual cycles not on hormone therapy.
* recently menopausal women (<3 years from final menstrual period) not on hormone therapy.

Premenopausal HypoE participants (women with functional hypothalamic amenorrhea) will be randomized to use either an estrogen patch or a placebo patch (no active medicine) for 12 weeks, followed by estrogen or placebo patch plus progesterone or placebo pills for 2 additional weeks. The investigators are looking to see if estrogen improves vascular and inflammation.

DETAILED DESCRIPTION:
Study Aims:

1. To test the hypothesis premenopausal HypoE (women with FHA) is associated with pre-clinical CVD as determined by reductions in vascular endothelial function.
2. To test the hypothesis premenopausal HypoE (women with FHA) is associated with increased immune-mediated inflammation.
3. To test the hypothesis whether estrogen replacement can reduce inflammation and improve vascular endothelial function in premenopausal HypoE women (women with FHA).

In a randomized, double-blind placebo-controlled trial in premenopausal HypoE women (women with FHA) the investigators will test 12 weeks of transdermal estradiol 0.1 mg/day patch or placebo followed by 2 weeks of estradiol plus progesterone 200mg (for endometrial safety) on vascular endothelial function and immune-mediated inflammation versus placebo. Patches will be applied by the participant to the lower abdomen twice weekly, alternating sides.

The investigators will be using non-invasive tests to measure vascular function to measures reactive hyperemic index (RHI) using peripheral arterial tonometry (PAT)

ELIGIBILITY:
Inclusion Criteria:

For premenopausal Hypo E and normal control women, inclusions include:

* Premenopausal currently not on hormone therapy,
* English speaking (for the purposes of complete psychosocial assessment)
* able to give informed consent
* a gynecological age (age since menarche) > 10 and < 25 years, and chronological age > 18 years
* Within 90-110% of ideal body weight as determined by the 1983 Metropolitan Height and weight table for women
* All participants with hypothalamic amenorrhea will be diagnosed based on exclusion of other etiologies for their amenorrhea, including pregnancy, thyroid dysfunction, hyperprolactinemia, premature ovarian insufficiency, and polycystic ovary disease

For recently menopausal women inclusions include:

* Follicle stimulating hormones (FSH) >30 and 12 months of amenorrhea, within 3 years of final menstrual period with natural menopausal not on hormone therapy
* English speaking
* Able to give informed consent
* Within 90-110% of ideal body weight

Exclusion Criteria:

For premenopausal Hypo E and normal control women exclusions include:

* Smoking
* Hypertension
* Hyperlipidemia
* Diabetes
* Medications including psychotropic or illicit drugs, medical, neurological
* Ophthalmologic disease except acuity problems
* Major Axis I disorder other than depression
* Pregnancy in the last 12 months and/or lactating in the last 6 months
* Current use of hormone contraceptive or any estrogen or progestin therapy

For HypoE women, exclusion criteria include:

- Allergy to adhesive or tape

For recently menopausal women exclusions also include:

* Previous or current use of hormone therapy, estrogen or progestin
* Surgical or chemotherapy induced menopause
* Premature ovarian failure

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chrisandra Shufelt, MD, Principal Investigator — Cedars-Sinai Medical Center; Noel Bairey-Merz, MD, Study Director — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Barbra Streisand Women's Heart Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shufelt CL, Saadedine M, Cook-Wiens G, Pisarska MD, Manson JE, Berga SL, Arditi M, Shah PK, Bairey Merz CN. Functional Hypothalamic Amenorrhea and Preclinical Cardiovascular Disease. J Clin Endocrinol Metab. 2023 Dec 21;109(1):e51-e57. doi: 10.1210/clinem/dgad498. PMID 37610989

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill
Started | 14 | 15
Completed | 12 | 12
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (6.7) | 25.1 (6.1) | 26.0 (6.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 8 | 18
  More than one race | 1 | 5 | 6
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21.7 (3.7) | 21.4 (3.1) | 21.5 (3.3)
Waist [Mean (Standard Deviation); unit: inches] | 27.1 (2.1) | 27.1 (3.7) | 27.1 (2.99)
Hip [Mean (Standard Deviation); unit: inches] | 34.0 (2.1) | 34.4 (3.7) | 34.2 (3.0)
Age at Menarche [Mean (Standard Deviation); unit: years] | 13.1 (1.8) | 12.9 (1.4) | 12.96 (1.6)
Serum Estradiol [Median (Inter-Quartile Range); unit: pg/mL] | 24 [12 to 42] | 30 [26 to 38] | 25 [18.5 to 35]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change of Reactive Hyperemia Index (RHI) by Peripheral Arterial Tonometry
Description: Change in PAT measured as reactive hyperemia index (RHI) from baseline to week 12 on treatment or placebo. Reactive hyperemia index (RHI) is the post-to-pre occlusion PAT signal ratio in the occluded arm, relative to the same ratio in the control arm, corrected for baseline vascular tone of the occluded arm calculated by taking the ratio of the pulse amplitude during the hyperemic phase (after a period of blood flow occlusion) to the baseline pulse amplitude. The values below <1.67 are abnormal and suggest impaired endothelial function or endothelial dysfunction.
Time Frame: Baseline, week 12 on trial
Population: Our results represent the change (delta) in RHI after 12 week of treatment vs placebo
Measure: Mean (Standard Deviation); unit: change of RHI
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill
Number analyzed (Participants) | 12 | 12
change of RHI | 0.20 (0.52) | 0.25 (0.64)

2. Secondary Outcome: Serum Inflammatory Markers
Description: Change in serum cortisol from baseline to week 12 on treatment or placebo
Time Frame: Change in serum cortisol from baseline to week 12 on treatment or placebo
Measure: Median (Inter-Quartile Range); unit: µg/dL
Groups:
- Transdermal Placebo Patch, Placebo Pill: Placebo Transdermal Patch, Placebo Pill for 12 weeks +/- 1 week. Placebos will be applied by the participant to the lower abdomen twice weekly, alternating sides.
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill
Number analyzed (Participants) | 12 | 12
µg/dL | -0.4 [-4.57 to 1.70] | 3.1 [0.2 to 5.96]

3. Secondary Outcome: Serum Estradiol Levels
Description: Week 12 serum estradiol levels
Time Frame: Serum estradiol levels after 12 week of treatment vs placebo
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill
Number analyzed (Participants) | 12 | 12
pg/mL | 108.0 [85.8 to 165.0] | 36.5 [16.7 to 51.2]

4. Secondary Outcome: Quality of Life (Questionnaire)
Description: Short-Form Health Survey 12 (SF-12) was reported as the mental component score (MCS) and physical component score (PCS). Each scale ranges from 0 to 100. For both PCS and MCS, higher values represent better outcomes, indicating superior physical or mental health, respectively. Lower scores suggest poorer outcomes in the respective domains. Scores above 50 for either PCS or MCS are generally considered above the population average for health-related quality of life, as the scales are often normed to a mean of 50 with a standard deviation of 10 in general population studies. Scores below 50 suggest below-average physical or mental health, with the degree of deviation providing further insight into the severity of physical or mental health challenges.
Time Frame: Change in quality of life scores after 12 week of treatment vs placebo
Population: Our results represent the change (delta) in quality of life scores after 12 week of treatment vs placebo for MCS and PCS.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Transdermal Placebo Patch, Placebo Pill: Placebo Transdermal Patch, Placebo Pill for 12 weeks
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill
Number analyzed (Participants) | 12 | 12
score on a scale
  SF12-PCS | 2.14 (7.97) | -0.45 (4.44)
  SF12-MCS | 1.83 (11.66) | 2.69 (5.99)

5. Secondary Outcome: Depression
Description: Patient Health Questionnaire (PHQ-9) total score ranges from 0 to 27. Each item is scored on a scale of 0 (not at all) to 3 (nearly every day), with higher scores indicating greater severity of depressive symptoms.
  Interpretation of Scores:
  * 0-4: Minimal or no depression
  * 5-9: Mild depression
  * 10-14: Moderate depression
  * 15-19: Moderately severe depression
  * 20-27: Severe depression
Time Frame: Change in PHQ-9 Scores after 12 week of treatment vs placebo
Population: Our results report the change (delta) in PHQ-9 after 12 week of estrogen treatment vs placebo.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill
Number analyzed (Participants) | 12 | 12
score on a scale | -0.67 (3.52) | -0.08 (2.09)

6. Secondary Outcome: Change in Insomnia Severity Index After 12 Week of Treatment vs Placebo
Description: Change in Insomnia Severity Index after 12 week of treatment vs placebo. Insomnia Severity Index (ISI) total score ranges from 0 to 28.
Time Frame: Insomnia score after 12 week of treatment vs placebo
Population: Our results report the change (delta) of the insomnia severity index after 12 week of estrogen treatment vs placebo
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill
Number analyzed (Participants) | 12 | 12
score on a scale | 8.0 (5.7) | 3.9 (4.0)

7. Secondary Outcome: Anxiety
Description: Overall Anxiety Severity and Impairment Scale (OASIS) total score ranges from 0 to 20, with each of the 5 items scored on a scale of 0 (no anxiety or impairment) to 4 (extreme anxiety or impairment). Higher scores indicate greater severity and functional impairment related to anxiety.
  The OASIS scores can be categorized as follows:
  * 0-4: Minimal or no anxiety
  * 5-9: Mild anxiety
  * 10-14: Moderate anxiety with some functional impairment
  * 15-20: Severe anxiety with significant functional impairment.
Time Frame: Change in Anxiety Scores after 12 week of treatment vs placebo
Population: Our results report the change (delta) in Anxiety Scores after 12 week of estrogen treatment vs placebo
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill
Number analyzed (Participants) | 12 | 12
score on a scale | -0.31 (3.3) | -0.54 (2.07)

8. Secondary Outcome: Stress
Description: Cohen Perceived Stress Scale (PSS) ranges from 0 to 40, with each of the 10 items scored on a scale of 0 (never) to 4 (very often). Higher scores reflect higher levels of perceived stress.
  The PSS scores can be categorized as follows:
  * 0-13: Low perceived stress
  * 14-26: Moderate perceived stress
  * 27-40: High perceived stress
Time Frame: Change in stress scores after 12 week of treatment vs placebo
Population: Our results indicate the change (delta) in stress scores after 12 week of estrogen treatment vs placebo.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill
Number analyzed (Participants) | 12 | 12
score on a scale | -0.49 (3.69) | -0.46 (3.41)

9. Secondary Outcome: Change in Serum Estradiol Levels
Description: Change from Baseline to week 12 serum estradiol levels
Time Frame: change in estradiol after 12 week of treatment vs placebo
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill
Number analyzed (Participants) | 12 | 12
pg/mL | 84 [44.3 to 144.8] | -4.7 [-14.6 to 4.25]

10. Secondary Outcome: Serum Inflammatory Markers
Description: Change in serum hsCRP from baseline to week 12 on treatment or placebo
Time Frame: Change in serum hsCRP from baseline to week 12 on treatment or placebo
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill
Number analyzed (Participants) | 12 | 12
mg/L | 0.0857 [0.017 to 0.174] | 0.0322 [-0.00021 to 0.172]

ADVERSE EVENTS:
Time Frame: For the length of the study enrollment, 14 weeks.
Arm/Group | 17Beta Estradiol, Progesterone | Transdermal Placebo Patch, Placebo Pill
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT03018366/Prot_SAP_000.pdf